CLINICAL TRIAL: NCT07374965
Title: A Prospective, Non-interventional, Single-Centre Study Assessing the Efficacy of a Holistic Upper Face Treatment With Botulinum Neurotoxin A
Status: Completed | Type: Observational
Sponsor: Yuvell (Other)
Collaborators: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: YUV-NIS-001
Record Dates: First submitted 2026-01-14; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Glabellar Lines; Forehead Lines; Crow's Feet; Canthal Lines
Keywords: botulinum toxin A; facial wrinkles; aesthetic medicine; forehead lines; crow's feet; glabellar lines; canthal lines
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Letybo® — Drug is used as part of routine clinical care. This observational study does not assign or modify treatment; it observes outcomes associated with drug use.
  Other Names: BoNT/A; botulinum toxin A; Letibotulinumtoxin A

SUMMARY:
The goal of this observational study is to learn about the safety, tolerability, and effectiveness of Letibotulinumtoxin A for the holistic treatment of the upper face in adults under 75 years old with moderate to severe upper facial lines, including glabellar lines, forehead lines, and lateral canthal lines.

The main questions it aims to answer are:

* Does Letibotulinumtoxin A safely and effectively reduce the severity of glabellar lines, forehead lines, and lateral canthal lines in adults under 75?
* How well is the treatment tolerated in everyday clinical practice?
* What is the patient satisfaction with holistic upper face treatment using Letibotulinumtoxin A?

Participants will:

* receive Letibotulinumtoxin A injections in the upper face, including glabellar lines, forehead lines, and lateral canthal lines.
* be observed and followed up to assess the severity of wrinkles, duration of effect, and patient satisfaction.
* report any adverse effects experienced during or after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at time of treatment.
* At least mild frown lines at maximum frown, mild dynamic forehead lines at maximum eyebrow elevation or mild crow's feet at maximum smile.
* Subject has a stable medical condition with no uncontrolled systemic disease.
* Willingness to participate in the routine follow - up after 2 weeks and 4 months and a signed informed consent form.

Exclusion Criteria:

* Pregnancy and breast feeding.
* Neuromuscular disease (e.g. myasthenia gravis, Eaton - Lambert syndrome).
* Known impairment of blood coagulation.
* Drooping eyelid.
* Known allergy to botulinum toxin or human albumin (blood protein).
* Presence of acute infection or inflammation at the proposed injection sites.
* Botulinumtoxin treatment in the upper face within the last 16 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting the clinic for such a treatment as part of routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a combined ≥ 1-point improvement in glabellar lines, forehead lines, and crow's feet severity at Week 2 | Week 2
  Proportion of subjects achieving a combined responder status, defined as an improvement of at least 1 point from baseline in all 3 treated facial regions at Week 2, as assessed by the investigator using the following validated photo-numeric scales:
  * Vertical glabellar lines assessed at maximum frowning using the Facial Wrinkle Scale (FWS), a scale ranging from 0 to 3, where higher scores indicate greater wrinkle severity.
  * Forehead lines assessed at maximum eyebrow elevation using the Croma Dynamic Forehead Line Assessment Scale (CDFLAS), a scale ranging from 1 to 5, where higher scores indicate greater wrinkle severity.
  * Crow's feet assessed at maximum smiling using the Croma Dynamic Crow's Feet Assessment Scale (CDCFAS), a scale ranging from 1 to 5, where higher scores indicate greater wrinkle severity.
  A subject is considered a responder only if the ≥ 1-point improvement criterion is met for all 3 scales simultaneously.

SECONDARY OUTCOMES:
Change in vectorial skin displacement at maximum frowning assessed by three-dimensional (3D) surface imaging | Week 2, Week 16
  Change from baseline in vectorial skin displacement at maximum frowning, measured at Week 2 and Week 16 using three-dimensional (3D) surface imaging technology.
  Vectorial skin displacement is quantified by comparing 3D facial surface images captured at baseline and follow-up visits to assess the magnitude and direction of skin movement during maximum frowning.
  Wrinkle severity at maximum frowning is additionally assessed by the investigator using the Facial Wrinkle Scale (FWS), a validated photo-numeric scale ranging from 0 to 3, where higher scores indicate greater wrinkle severity, to provide clinical context for the imaging-based measurements.
Change in vectorial skin displacement during maximum frontalis muscle contraction assessed by three-dimensional (3D) surface imaging | Week 2, Week 16
  Change from baseline in vectorial skin displacement during maximum frontalis muscle contraction, assessed at Week 2 and Week 16 using three-dimensional (3D) surface imaging technology.
  Vectorial skin displacement is quantified by comparing 3D facial surface images obtained at baseline and follow-up visits to evaluate the magnitude and direction of skin movement over the forehead region during maximum frontalis muscle contraction.
  Forehead wrinkle severity during maximum contraction is additionally assessed by the investigator using the Croma Dynamic Forehead Line Assessment Scale (CDFLAS), a validated photo-numeric scale ranging from 1 to 5, where higher scores indicate greater wrinkle severity, to provide clinical context to the imaging-based measurements.
Change in vectorial skin displacement during maximum orbicularis oculi muscle contraction assessed by three-dimensional (3D) surface imaging | Week 2, Week 16
  Change from baseline in vectorial skin displacement during maximum orbicularis oculi muscle contraction, assessed at Week 2 and Week 16 using three-dimensional (3D) surface imaging technology.
  Vectorial skin displacement is quantified by comparing 3D facial surface images captured at baseline and follow-up visits to evaluate the magnitude and direction of skin movement in the periocular (crow's feet) region during maximum orbicularis oculi muscle contraction.
  Wrinkle severity of the crow's feet during maximum contraction is additionally assessed by the investigator using the Croma Dynamic Crow's Feet Assessment Scale (CDCFAS), a validated photo-numeric scale ranging from 1 to 5, where higher scores indicate greater wrinkle severity, to provide clinical context for the imaging-based displacement measurements.
Percentage of subjects requiring a touch-up at Week 2 | Week 2
  Percentage of subjects who, in the opinion of the investigator, required a touch-up treatment at the Week 2 visit to optimize the treatment outcome.
  The need for a touch-up is determined by the investigator based on clinical assessment.
Patient satisfaction with treatment assessed using a clinic-internal patient satisfaction questionnaire | Week 16
  Patient satisfaction with the treatment as assessed by participants using the clinic-internal questionnaire titled "Patient Satisfaction Questionnaire".
  The questionnaire consists of 5 questions evaluating the participant's overall satisfaction with the treatment outcome. Each item is rated on a numeric ordinal scale from 1 to 5, where lower scores indicate higher patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Duschek, Priv.-Doz., PhD, Principal Investigator — Yuvell
Locations (1):
- YUVELL, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided